CLINICAL TRIAL: NCT01979614
Title: A Multicenter, Double Blind, Randomized, Parallel Group, Placebo-controlled Study to Evaluate the Effects of Intravenous Serelaxin Infusion on Micro- and Macrovascular Function in Patients With Coronary Artery Disease
Brief Title: Study of the Vascular Effects of Serelaxin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRLX030A2203; 2012-001945-42 (EudraCT Number)
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — serelaxin protein, human; Relaxin

STUDY DESIGN:
Intervention Model Description: double blind, randomized, parallel group, placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serelaxin (Experimental): Serelaxin was administered at a dose of 30 μg/kg/24h by intravenous infusion for 48 hours
  Interventions: Drug: Serelaxin
- Placebo (Placebo Comparator): Placebo was administered by intravenous infusion for 48 hours
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Serelaxin — Serelaxin solution diluted in 5% glucose volume/volume (v/v) solution
  Other Names: RLX030, relaxin
  Arms: Serelaxin
Other: Placebo — 5% v/v glucose solution
  Arms: Placebo

SUMMARY:
This was a mechanistic study in patients with coronary artery disease on the effects of Serelaxin on micro- and macrovascular function.

DETAILED DESCRIPTION:
double blind, randomized, parallel group, placebo controlled study

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years of age, with body weight <160 kg.
* Patients with proven obstructive coronary artery disease, determined either by functional (e.g. treadmill testing) or non-invasive clinical imaging assessments (e.g. stress-echo, PET or SPECT myocardial perfusion), or invasive coronary angiography or by CT coronary angiography at any point in time in patients with or without mild left ventricular systolic dysfunction (LVSD)

Exclusion Criteria:

* Previous treatment with serelaxin (also known as: RLX030, relaxin)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of study treatment.
* Current or planned dialysis.
* Impaired renal function during screening defined as an estimated glomerular filtration rate (eGFR) at screening and prior to treatment of <30 mL/min/1.73 m2, calculated using the simplified Modification of Diet in Renal Disease (sMDRD) equation due to potential issue with administration of GdDTPA used as the MRI contrast agent.
* Sick-Sinus-Syndrome
* Current or history of pulmonary edema, including suspected sepsis.
* restrictive, or constrictive cardiomyopathy (does not include restrictive mitral filling patterns seen on Doppler echocardiographic assessments of diastolic function)
* Known significant valvular disease (including any of the following: severe aortic stenosis [AVA < 1.0 or peak gradient > 50 on prior or current echocardiogram], severe aortic regurgitation, or severe mitral stenosis).
* Clinical diagnosis of acute coronary syndrome (ACS) including unstable angina within 30 days prior to screening as determined by both clinical and enzymatic criteria
* Troponin elevation and dynamics indicative of ACS at any time between screening and randomization.
* Previous myocardial infarction within 3 months of screening
* History of Coronary Artery Bypass Graft (CABG) surgery
* Heart failure due to significant arrhythmias (including any of the following: ventricular tachycardia, bradyarrhythmias with ventricular rate < 45 beats per minute or any second or third degree AV block or atrial fibrillation/flutter with ventricular response of > 120 beats per minute)
* Any surgical or medical condition which in the opinion of the investigator may place the patient at higher risk from his/her participation in the study (e.g., history of poor tolerance of adenosine or 3 vessel coronary disease)
* Acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy (does not include restrictive mitral filling patterns seen on Doppler echocardiographic assessments of diastolic function).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2016-08-17 (Actual); Study Completion 2016-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United Kingdom (3):
  - Novartis Investigative Site, Clydebank, West Dumbartonshire
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Leicester

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the total 63 participants screened, 62 were randomized. 4 of the randomized participants did not receive study drug, and 58 did receive study drug
Pre-assignment Details: Of the 58 participants in the safety analysis set, 56 completed the treatment and follow-up period as planned (i.e. Day 30 and Day 180).
Period: Overall Study
Arm/Group | Serelaxin | Placebo
Started | 30 | 28
Safety Analysis Set | 30 | 28
PK Analysis Set | 30 | 0
PD Analysis Set | 25 | 26
Completed | 29 | 27
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Serelaxin | Placebo | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (6.42) | 60.1 (7.05) | 61.4 (6.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Statistical Analysis of Change From Baseline to Day 3 in Myocardial Perfusion Endpoints Compared With Mid Perfusion Reserve Index Using ANCOVA End Points
Description: Global MPRI (Myocardial Perfusion Reserve Index) is defined as ratio between mean global myocardial blood flow values at rest and during adenosine stress with Mid Perfusion Reserve Index or Midl PRI (Mid Perfusion Reserve Index) which is defined as ratio between mid myocardial blood flow values at rest and during adenosine stress
Time Frame: baseline to Day 3
Population: The Pharmacodynamic (PD) analysis set included all patients with available PD data who received any study drug and experienced no protocol deviations with relevant impact on PD data.
  Participants who did not receive study drug as per study protocol, i.e. a reduced infusion rate, were excluded from this analysis
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Serelaxin | Placebo
Number analyzed (Participants) | 22 | 25
ratio
  Global Myocardial Perfusion Reserve Index (MPRI) | -0.244 [-0.454 to -0.035] | -0.133 [-0.329 to -0.064]
  Mid Perfusion Reserve Index | -0.264 [-0.519 to -0.010] | -0.075 [-0.313 to 0.164]
Statistical Analysis 1: Comparison: Serelaxin vs Placebo; SAP for Global Myocardial Perfusion Reserve Index (MPRI); Test type: Superiority or Other; p = 0.438, ANCOVA; Standard Error = -0.1116, 95% CI 2-sided [-0.399 to 0.176]

2. Secondary Outcome: Change From Baseline in Aortic Distensibility Measured by MRI
Description: Measurements of arterial stiffness from cardiac MRI - Mean (SD) [n]
  Aortic distensibility was assessed by MRI and pulse wave velocity using the SphygmoCor device.
  (mmHg-1)
Time Frame: At pre-dose on Day 1 (baseline) until Day 180 after the start of drug infusion
Population: PD Analysis Set
Measure: Mean (Standard Deviation); unit: mmHg-1
Arm/Group | Serelaxin | Placebo
Number analyzed (Participants) | 25 | 26
mmHg-1
  Ascending Aorta Distensibility, Day 0: number analyzed (Participants) | 24 | 22
  Ascending Aorta Distensibility, Day 0 | 0.0017 (0.00158) | 0.0014 (0.00192)
  Ascending Aorta Distensibility, Day 47: number analyzed (Participants) | 23 | 22
  Ascending Aorta Distensibility, Day 47 | 0.0015 (0.00124) | 0.0015 (0.00134)
  Descending Aorta Distensibility, Day 0: number analyzed (Participants) | 24 | 21
  Descending Aorta Distensibility, Day 0 | 0.0023 (0.00146) | 0.0019 (0.00221)
  Descending Aorta Distensibility, Day 47: number analyzed (Participants) | 23 | 22
  Descending Aorta Distensibility, Day 47 | 0.0023 (0.00118) | 0.0023 (0.00142)

3. Secondary Outcome: Change From Baseline in Aortic Velocity
Description: Summary table for measurements of arterial velocity from cardiac MRI - Mean (SD) [n]
  Aortic distensibility was assessed by MRI and pulse wave velocity using the SphygmoCor device
Time Frame: At pre-dose on Day 1 (baseline) until Day 180 after the start of drug infusion
Population: PD Analysis Set
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Serelaxin | Placebo
Number analyzed (Participants) | 25 | 26
cm/s
  Peak Flow Velocity (cm/s), Day 0 (n=24, 24): number analyzed (Participants) | 24 | 24
  Peak Flow Velocity (cm/s), Day 0 (n=24, 24) | 127.981 (60.7571) | 106.557 (38.9573)
  Peak Flow Velocity (cm/s), Day 47 (n=23, 25): number analyzed (Participants) | 23 | 25
  Peak Flow Velocity (cm/s), Day 47 (n=23, 25) | 127.981 (60.7571) | 106.557 (38.9573)

4. Secondary Outcome: Change From Baseline in Augmentation Index Measured From Sphygmocor Device
Description: Summary of values and change from baseline in augmentation index by time and treatment
  The change from baseline in Augmentation Index was analyzed using a repeated measures analysis of covariance including treatment, time, treatment by time, baseline by time interactions and baseline as fixed factors with an unstructured variance-covariance matrixStatistical analysis of change from baseline in augmentation index using repeated measures Analysis of Covariance
Time Frame: Day1, Day 2, Day 3, Day 30 and Day 180 after the start of infusion
Population: PD Analysis Set For analysis of change from baseline, only subjects with results at both baseline and post-baseline could be included
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Serelaxin | Placebo
Number analyzed (Participants) | 25 | 26
ratio
  DAY 1, 2h (n=23,25): number analyzed (Participants) | 23 | 25
  DAY 1, 2h (n=23,25) | -4.12 (11.441) | -2.48 (11.560)
  DAY 1, 6h (n=24,26): number analyzed (Participants) | 24 | 26
  DAY 1, 6h (n=24,26) | -2.99 (9.066) | -0.58 (9.551)
  DAY 2, 24h (n=24,25): number analyzed (Participants) | 24 | 25
  DAY 2, 24h (n=24,25) | -0.82 (8.173) | 0.22 (9.906)
  DAY 3, 47h (n=23,25): number analyzed (Participants) | 23 | 25
  DAY 3, 47h (n=23,25) | 3.51 (10.608) | 0.22 (12.057)
  DAY 3, 50h (n=22, 24): number analyzed (Participants) | 22 | 24
  DAY 3, 50h (n=22, 24) | -0.67 (13.034) | -3.81 (9.397)
  DAY 3, 54h (n=22,25): number analyzed (Participants) | 22 | 25
  DAY 3, 54h (n=22,25) | -1.37 (12.253) | -0.48 (11.748)
  DAY 30 (n=25, 26) | -0.83 (11.462) | 0.58 (12.124)
  DAY 180 (n=24,25) end of study: number analyzed (Participants) | 24 | 25
  DAY 180 (n=24,25) end of study | 0.24 (6.885) | 0.54 (11.795)

5. Secondary Outcome: Statistical Analysis of Change From Baseline in Augmentation Index Using Repeated Measures Analysis of Covariance
Description: The change from baseline in Augmentation Index was analyzed using a repeated measures analysis of covariance including treatment, time, treatment by time, baseline by time interactions and baseline as fixed factors with an unstructured variance-covariance matrixStatistical analysis of change from baseline in augmentation index using repeated measures Analysis of Covariance
  For analysis of change from baseline, only subjects with results at both baseline and post-baseline could be included
  The augmentation index is a ratio calculated from the blood pressure waveform, it is a measure of wave reflection and arterial stiffness. Augmentation index is commonly accepted as a measure of the enhancement (augmentation) of central aortic pressure by a reflected pulse wave
Time Frame: Day1, Day 2, Day 3, Day 30 and Day 180 after the start of infusion
Population: PD Analysis Set
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Serelaxin | Placebo
Number analyzed (Participants) | 25 | 26
ratio
  DAY 1, 2h (n=23,25): number analyzed (Participants) | 23 | 25
  DAY 1, 2h (n=23,25) | -4.088 [-7.967 to -0.210] | -1.970 [-5.693 to 1.753]
  DAY 1, 6h (n=24,26): number analyzed (Participants) | 24 | 26
  DAY 1, 6h (n=24,26) | -3.277 [-6.129 to -0.425] | -0.394 [-3.139 to 2.352]
  DAY 2, 24h (n=24,25): number analyzed (Participants) | 24 | 25
  DAY 2, 24h (n=24,25) | -0.774 [-4.016 to 2.469] | 0.070 [-3.108 to 3.247]
  DAY 3, 47h (n=23,25): number analyzed (Participants) | 23 | 25
  DAY 3, 47h (n=23,25) | 3.488 [-0.470 to 7.445] | 0.035 [-3.778 to 3.849]
  DAY 3, 50h (n=22, 24): number analyzed (Participants) | 22 | 24
  DAY 3, 50h (n=22, 24) | -0.764 [-5.208 to 3.680] | -4.015 [-8.273 to 0.243]
  DAY 3, 54h (n=22,25): number analyzed (Participants) | 22 | 25
  DAY 3, 54h (n=22,25) | -1.737 [-5.915 to 2.440] | -0.753 [-4.689 to 3.182]
  DAY 30 (n=25, 26) | -0.979 [-4.912 to 2.954] | 0.776 [-3.081 to 4.633]
  DAY 180 (n=24,25) end of study: number analyzed (Participants) | 24 | 25
  DAY 180 (n=24,25) end of study | 0.234 [-3.066 to 3.535] | 0.284 [-2.950 to 3.518]

6. Secondary Outcome: Change From Baseline in Pulse Wave Velocity Measured From Carotid-femoral Pulse Wave Analysis
Description: Pulse wave velocity was assessed by the SphygmoCor device
Time Frame: Day1, Day 2, Day 3, Day 30 and Day 180 after the start of infusion
Population: The Pharmacodynamic (PD) analysis set included all patients with available PD data who received any study drug and experienced no protocol deviations with relevant impact on PD data. Any patients who had a reduced flow rate of infusion were excluded from this analysis
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Serelaxin | Placebo
Number analyzed (Participants) | 25 | 26
meters/second
  DAY 1, 0hrs (n=25,26) | 7.453 (2.0541) | 8.166 (1.9515)
  DAY 2, 24hrs (n=19,24): number analyzed (Participants) | 19 | 24
  DAY 2, 24hrs (n=19,24) | 7.051 (1.8790) | 7.677 (2.1361)
  DAY 3, 47hrs (n=22,23): number analyzed (Participants) | 22 | 23
  DAY 3, 47hrs (n=22,23) | 7.195 (1.9164) | 8.264 (2.4964)
  DAY 30, 0hrs (n=23, 24): number analyzed (Participants) | 23 | 24
  DAY 30, 0hrs (n=23, 24) | 7.989 (1.8151) | 8.463 (2.4437)
  DAY 3, 47hrs (n=23,25): number analyzed (Participants) | 23 | 25
  DAY 3, 47hrs (n=23,25) | 29.57 (9.751) | 26.04 (10.039)
  DAY 180 EOS (n=23,24): number analyzed (Participants) | 23 | 24
  DAY 180 EOS (n=23,24) | 8.335 (2.1087) | 8.844 (2.1739)

7. Secondary Outcome: Serum Concentration of Serelaxin
Description: Summary statistics of serelaxin serum PK concentrations
  Blood samples were taken to measure serelaxin concentration
Time Frame: Day1, Day 2, Day 3 and Day 30 after the start of infusion
Population: Pharmacokinetic Analysis Set
  The PK analysis set includes all participants with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, who received any study drug and experienced no protocol deviations with relevant impact on PK data
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Serelaxin
Number analyzed (Participants) | 30
pg/mL
  DAY 1, 0hrs (n=30) | 0.637 (3.49)
  DAY 2, 24hrs, (n=26): number analyzed (Participants) | 26
  DAY 2, 24hrs, (n=26) | 27600 (79000)
  DAY 3, 48hrs (n=22): number analyzed (Participants) | 22
  DAY 3, 48hrs (n=22) | 26300 (48000)
  DAY 3, 50 hrs (n=21): number analyzed (Participants) | 21
  DAY 3, 50 hrs (n=21) | 7940 (8450)
  DAY 3, 54hrs, (n=22): number analyzed (Participants) | 22
  DAY 3, 54hrs, (n=22) | 3960 (3140)
  DAY 30 (n=30) | 0.00 (0.00)

8. Secondary Outcome: Serum Concentration of Antibodies to Serelaxin
Description: Frequency and percentage of anti-Serelaxin antibodies
  Blood samples were taken to measure antibodies to serelaxin concentration at Pre-dose on Day 1, and at Day 30 after the start of the 48h drug infusion
Time Frame: From pre-dose on Day 1 until Day 30 after the start of drug infusion
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Serelaxin | Placebo
Number analyzed (Participants) | 30 | 28
percentage of participants
  DAY 1 NEGATIVE | 100 | 100
  DAY 1 POSITIVE | 0 | 0
  DAY 30 NEGATIVE | 100 | 100
  DAY 30 POSITIVE | 0 | 0

9. Secondary Outcome: Systemic Clearance of Serelaxin
Description: Systemic clearance was estimated using the rate of serelaxin infusion and the steady state concentration
Time Frame: From pre-dose on Day 1 until 48h after the start of drug infusion
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | Serelaxin
Number analyzed (Participants) | 22
mL/hr/kg | 107 (80.6)

ADVERSE EVENTS:
Time Frame: Day 180
Groups:
- Serelaxin: Serelaxin
- Placebo: Placebo
Arm/Group | Serelaxin | Placebo
Serious Adverse Events (participants affected / at risk) | 5/30 | 7/28
Other Adverse Events (participants affected / at risk) | 16/30 | 18/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Serelaxin (N=30) | Placebo (N=28)
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Type IV hypersensitivity reaction (Immune system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Serelaxin (N=30) | Placebo (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 2
Extrasystoles (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Feeling cold (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Amylase increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood sodium decreased (Investigations) | 0 | 1
Electrocardiogram Q wave abnormal (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0
Haematocrit decreased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 2 | 2
Lipase increased (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
QRS axis abnormal (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 2 | 4
Presyncope (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.